CLINICAL TRIAL: NCT04949425
Title: An Open-label, Non-randomised, Multicentre Study to Allow Continued Access to and Assess the Safety and Tolerability of Adavosertib for Patients With Advanced Solid Tumours Enrolled in Adavosertib Clinical Pharmacology Studies
Brief Title: A Study to Assess the Safety and Tolerability of Adavosertib for Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated because the clinical development programme for Adavosertib has been discontinued
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D601HC00009
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumours
Keywords: Advanced Solid Tumours; Continued Access; Parent Studies
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with advanced solid tumours (Experimental): Patients with advanced solid tumours will receive Adavosertib once daily for 5 days followed by 2 days off for 2 weeks out of a 21-day cycle.
  Interventions: Drug: Adavosertib

INTERVENTIONS:
Drug: Adavosertib — Patients will receive Adavosertib orally.
  Other Names: AZD1775

SUMMARY:
The purpose of this study is to allow continued adavosertib treatment of patients with advanced solid tumours participating in the adavosertib clinical pharmacology studies and to assess the continued safety and tolerability of adavosertib for patients enrolled in adavosertib clinical pharmacology studies (hereafter referred to as the 'parent studies') who continue to use the therapy

DETAILED DESCRIPTION:
Patients will be screened within 14 days of Day 1 of the treatment period. During screening, patients will undergo an appropriate washout period after the last dose of adavosertib in the parent clinical pharmacology study before receiving the first dose of adavosertib in this study.

Patients will continue to receive adavosertib as long as they are benefiting from treatment in the investigator's opinion and do not meet any other discontinuation criteria.

The number of patients who enroll is dependent on the number of patients who complete the parent studies, and who tolerate adavosertib in the parent study.

The anticipated total duration of the study is approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
2. Participant has completed one of the parent adavosertib clinical pharmacology studies (i.e., D601HC00004, D601HC00006) and is suitable for continued treatment with adavosertib.
3. Eastern Cooperative Oncology Group performance status score of 0 to 1.
4. Life expectancy ≥ 12 weeks.
5. Participants must have normal organ and marrow function at baseline, within 7 days prior to study drug administration.
6. Males and females of childbearing potential who agree to use contraceptive measures should be consistent with clinical study protocol.

Exclusion Criteria:

1. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade > 2) caused by previous anticancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy.
2. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of adavosertib.
3. Any significant cardiac diseases currently or within the last 6 months such as:

   1. unstable angina pectoris
   2. acute myocardial infarction, congestive heart failure
   3. conduction abnormality not controlled with pacemaker or medication
   4. significant ventricular or supraventricular arrhythmias
4. Any of the following: History or current evidence of congenital long QT syndrome; concomitant medications known to prolong QT interval or history of medication-related QT prolongation.
5. Known to have tested positive for human immunodeficiency virus or active tuberculosis infection.
6. Known active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening.
7. Any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, active infections, and active bleeding diseases) which prohibit participating in the study.
8. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.
9. Use of an anti-cancer treatment drug ≤ 21 days (≤ 6 weeks for nitroureas or mitomycin C) or use of an investigational product within 5 half-lives prior to the first dose of adavosertib.
10. Patient uses drugs that are sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or are moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks or 5 halflives (whichever is longer) prior to Day 1 of dosing.
11. Receipt of live virus and live bacterial vaccines whilst the patient is receiving the study intervention and during the 30-day follow-up period. Inactivated vaccines are permitted.
12. Currently pregnant (confirmed with positive pregnancy test) or breast feeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with serious and non-serious adverse events | From screening to safety follow-up (30 days after last dose)
  Assessment of the safety and tolerability of adavosertib following oral dosing of the capsule formulation in patients with advanced solid tumours

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Dallas, Texas, United States
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the
  Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home